CLINICAL TRIAL: NCT00558233
Title: Overcoming Literacy Barriers in Colorectal Cancer Screening
Brief Title: Effectiveness Study of a Computer-Based Colorectal Cancer Screening Decision Aid
Acronym: InfoPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Cancer Society, Inc. (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CCCDA-05-162-01
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Cancer; Health Literacy
Keywords: Colorectal cancer; Screening; Health literacy; Patient education; Computer assisted instruction
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: CHOICE decision aid
- Placebo group (Placebo Comparator)
  Interventions: Behavioral: YourMeds patient education program

INTERVENTIONS:
Behavioral: CHOICE decision aid — computer-based patient decision aid about colorectal cancer screening delivered immediately before a healthcare provider visit
  Other Names: CHOICE
  Arms: Intervention group
Behavioral: YourMeds patient education program — computer-based patient education program about prescription drug safety seen immediately before a healthcare provider visit
  Other Names: YourMeds
  Arms: Placebo group

SUMMARY:
The purpose of this study is to determine whether a multimedia educational computer program can increase colorectal cancer screening rates in low and adequate literacy patients.

DETAILED DESCRIPTION:
Results will be stratified by low/marginal and adequate literacy as determined by the Rapid Estimate of Adult Literacy in Medicine instrument.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Scheduled to see an internal medicine provider
* No recent colorectal cancer screening

Exclusion Criteria:

* Personal history of colorectal cancer
* Family history of colorectal cancer
* Blood seen in stools within last month
* Obvious cognitive or physical impairment that would prevent participation

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2007-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Receipt of colorectal cancer screening | 24 weeks

SECONDARY OUTCOMES:
Change in participants' readiness to be screened (Stage of Change) | Day 1
Self-reported intent to discuss colorectal cancer screening with healthcare provider | Day 1
Provider ordering a colorectal cancer screening test | Day 1
Participant completion of computer program without assistance | Day 1
Participant acceptance of computer program | Day 1
Number of polyps and cancers found by screening tests performed | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David P Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Baptist Medical Center; Downtown Health Plaza, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Miller DP Jr, Spangler JG, Case LD, Goff DC Jr, Singh S, Pignone MP. Effectiveness of a web-based colorectal cancer screening patient decision aid: a randomized controlled trial in a mixed-literacy population. Am J Prev Med. 2011 Jun;40(6):608-15. doi: 10.1016/j.amepre.2011.02.019. PMID 21565651